CLINICAL TRIAL: NCT06561932
Title: A Feasibility Study Implant of the WiSE® CRT System With an Intracardiac Pacemaker to Achieve Totally Leadless CRT
Acronym: TLC-AU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: EBR Systems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSP-10002
Record Dates: First submitted 2024-08-08; First posted 2024-08-20 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Single-arm, prospective, multicenter, observational study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-arm, prospective, multicenter, observational study. (Experimental): .WiSE System therapy ON with Guideline Directed Medical Therapy
  Interventions: Device: WiSE CRT System

INTERVENTIONS:
Device: WiSE CRT System — The WiSE CRT System is an implantable cardiac system to provide left ventricular (LV) pacing stimulation in conjunction with a co-implanted system that provides right ventricular (RV) stimulation. In combination, the devices deliver biventricular (BiV) pacing.

SUMMARY:
Assess the safety and efficacy of the co-implantation of the WiSE CRT System with an intracardiac pacemaker to provide totally leadless CRT.

DETAILED DESCRIPTION:
The WiSE CRT System is an implantable cardiac system to provide left ventricular (LV) pacing stimulation in conjunction with a co-implanted system that provides right ventricular (RV) stimulation. In combination, the devices deliver biventricular (BiV) pacing.

Single-arm, prospective, multicenter, observational study.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a class I or IIa (1) or (2) indication for implantation of a CRT device according to current available guidelines 1,2,4 (with additional QRS criteria on Class IIa (1)):

  * Class I: NYHA II, III, IV, EF ≤ 35%, LBBB, QRS ≥ 150 ms
  * Class IIa (1): NYHA II, III, IV, EF ≤ 35%, LBBB, QRS ≥ 130 to < 150 ms
  * Class IIa (2): NYHA II, III, IV, EF ≤ 35%, non-LBBB, QRS ≥ 150 ms
* Patient or legally authorized representative can provide written authorization and/or consent per institution requirements
* Male or Female, aged 22 years or above
* Meets criteria for one of the two patient groups

  * Group A: De novo totally leadless CRT implant in whom the physician believes a totally leadless approach would be beneficial (e.g., wish to avoid lifelong transvenous lead implant, anatomical constraints, history of device infection).

    * Patients with symptomatic AF and an uncontrolled heart rate who are candidates for AV node ablation (irrespective of QRS duration and LVEF), and in whom the physician believes a leadless pacing approach would be beneficial.
    * Patients with high degree AV block who have an indication for permanent pacing (with a LVEF ≤ 50%), are expected to require ventricular pacing more than 40% of the time, and in whom the physician believes a leadless approach would be beneficial.
  * Group B: Upgrade chronic intracardiac pacemaker to CRT

    * Patients with existing intracardiac pacemakers with greater than 20% RV pacing, who have developed symptomatic HF.

Exclusion Criteria:

* Patient who is or is expected to be inaccessible for follow-up visits
* Female participant who is pregnant, lactating, or planning pregnancy during the course of the study
* Inability to comply with the study follow-up or other study requirements
* History of chronic alcohol/ drug abuse and currently using alcohol/ drugs
* Non-ambulatory (or unstable) NYHA class 4
* Life expectancy less than 12 months
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.
* Patient who is enrolled in another clinical study that could confound the results of this study (Note: patients enrolled in complementary study are eligible for enrolment)

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-18 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Device and procedure related complications. | 1 month and 6 months
  Primary Safety
Bi-Ventricular capture on 12 lead EKG | 1 month and 6 months
  Performance

SECONDARY OUTCOMES:
Change in ejection fraction (EF) from Baseline | 6 months
  Secondary efficacy 1
Change in in left ventricular end systolic volume (LVESV) | 6 months
  Secondary efficacy 2
Change in NYHA class | 6 months
  Secondary efficacy 3
Change in Six-minute walk test | 6 months
  Secondary efficacy 4

CONTACTS AND LOCATIONS:
Overall Officials: Paul Gould, Prof, Principal Investigator — Princess Alexandra Hospital
Locations (4):
- Australia (4):
  - Patients of Sunshine Coast University Hospital, Birtinya, Queensland
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Patients of Gold Coast University Hospital, Southport, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland